CLINICAL TRIAL: NCT03040193
Title: Nebulized Lignocaine for Topical Airway Anesthesia During Flexible Bronchoscopy: A Randomized Controlled Trial
Acronym: NEBULA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr Karan Madan MD, DM Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Ref.No.IEC-594/05.01.2017
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Bronchopulmonary Disease
Keywords: Lignocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized Lignocaine (Experimental): 4% Lignocaine administered as nebulization for topical anaesthesia during bronchoscopy procedure
  Interventions: Drug: Lignocaine Nebulization
- Nebulized Saline (Placebo Comparator): Normal Saline administered as nebulization for topical anaesthesia during bronchoscopy procedure
  Interventions: Drug: Saline Nebulization

INTERVENTIONS:
Drug: Lignocaine Nebulization — 4% Lignocaine delivered via Nebulization
  Arms: Nebulized Lignocaine
Drug: Saline Nebulization — Normal Saline Delivered via Nebulization
  Arms: Nebulized Saline

SUMMARY:
Flexible bronchoscopy is one of the most widely performed procedures for diagnosis of various bronchopulmonary diseases. Most patients tolerate the procedure well although cough is often reported as a distressing symptom. It is likely that the acceptance of bronchoscopy would be significantly improved with control of cough. Use of sedation during bronchoscopy has been reported to improve procedure tolerance. However, awake(no sedation) bronchoscopy is routinely performed at many centres including ours.

Topical lignocaine is administered during bronchoscopy for local anaesthesia. There is limited literature on the efficacy of lignocaine delivered with the nebulized route during awake flexible bronchoscopy. This study would help to determine the utility of nebulized lignocaine in airway anaesthesia during flexible bronchoscopy.

DETAILED DESCRIPTION:
For all patients meeting the inclusion criteria, the demographic profile including age, sex, weight, smoking history and the type of procedures performed during bronchoscopy shall be recorded. A written informed consent will be obtained from all participants. The patients who undergo flexible bronchoscopy would be randomised in a one is to one ratio either to nebulized lignocaine (4%) or saline (placebo) nebulization group. Prior to the bronchoscopy blood pressure, pulse rate, respiratory rate and pulse oximetry saturation will be recorded at the baseline Patients in both the groups shall be prepared in a similar fashion except for the nebulized lignocaine. Patient, Operator, outcome assessor will be blinded to the allocation.

During the procedure, 1.5ml aliquots of 1% lignocaine will be delivered through the bronchoscope using spray-as-you go technique. The patients would be monitored for any adverse effects throughout the procedure. The bronchoscopist doing the procedure will be provided 2 VAS charts to mark the severity of cough and overall procedure satisfaction.

Post procedure, patients will record the pain experienced while undergoing the procedure on the faces pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult (Age > 18 years) patients undergoing diagnostic or therapeutic flexible bronchoscopy

Exclusion Criteria:

1. Pregnancy
2. Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3
3. Bronchoscopy done through endotracheal or tracheostomy tube
4. Not willing to provide informed consent.
5. Patient requiring sedation for flexible bronchoscopy
6. Patients with known allergy to lignocaine -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Operator rated overall procedure satisfaction VAS | At study completion approx. 12 months
Operator rated cough VAS | At study completion approx. 12 months

SECONDARY OUTCOMES:
Total dose of Lignocaine administered (mg) | At study completion approx. 12 months
Number of patients receiving dose >8.2mg/Kg | At study completion approx. 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD, DM, Study Chair — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided